CLINICAL TRIAL: NCT05740345
Title: Management of Hyperglycemia in INOCA Patients
Brief Title: New Approaches to INOCA
Status: Completed | Type: Observational
Sponsor: Pasquale Mone (Other)
Responsible Party: Sponsor-Investigator, Pasquale Mone, Principal Investigator, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Other Study IDs: Campania Nord 2
Record Dates: First submitted 2023-01-30; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: New Approaches in INOCA
Keywords: INOCA; Hyperglycemia; Metformin; Endothelial Dysfunction; PCI
MeSH Terms: conditions — Hyperglycemia | interventions — Metformin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hyperglycemia/Normoglycemia
- Treated/No treated
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin
  Groups: Treated/No treated

SUMMARY:
Ischemia with non-obstructive coronary arteries (INOCA) is common in patients with angina. INOCA has been associated with an increased risk of death, myocardial infarction, and stroke, particularly in symptomatic subjects. Previous investigations have evidenced the key role of poor glycemic control and diabetes in coronary microvascular dysfunction. Metformin is an old oral antidiabetic drug which is currently used to achieve glycemic control.

DETAILED DESCRIPTION:
Ischemia with non-obstructive coronary arteries (INOCA) is common in patients with angina. INOCA has been associated with an increased risk of death, myocardial infarction, and stroke, particularly in symptomatic subjects. Coronary microvascular dysfunction, triggering structural remodeling and vasomotor disorders of coronary arterioles, is currently one of the leading hypotheses to explain INOCA pathophysiology. Previous investigations have evidenced the key role of poor glycemic control and diabetes in coronary microvascular dysfunction. Metformin is an old oral antidiabetic drug which is currently used to achieve glycemic control. Also, previous reports evidenced that metformin improves endothelial dysfunction. Nowadays, it is used in prediabetic patients too. In this scenario, we evaluated the role of metformin in reducing the risk of re-hospitalization in INOCA.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* diagnosis of INOCA;
* availability to participate in the study

Exclusion Criteria:

* cancer;
* atrial fibrillation or left bundle branch block;
* previous acute coronary syndrome (ACS) or cardiac revascularization; -pregnancy;
* severe heart valve disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: INOCA with Hyperglycemia
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Risk of Re-Hospitalization | 2016-2021
  Risk of Re-Hospitalization. The primary outcome measure will be the risk of re-hospitalization; to assess this outcome, we will assess the actual number of re-hospitalization events for each patients.

SECONDARY OUTCOMES:
MACE | 2016-2021
  Major adverse cardiovascular event (MACE):
  Acute myocardial infarction or acute coronary syndrome, stroke, cardiovascular death, all-cause death

IPD SHARING:
Plan to Share IPD: Undecided